CLINICAL TRIAL: NCT00475488
Title: Randomised Trial of Graft Patency and Clinical Outcomes, Comparing Radial Artery With Either the Right Internal Thoracic Artery or Saphenous Vein
Brief Title: Radial Artery Patency and Clinical Outcomes Trial
Acronym: RAPCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Austin Health (Other Government)
Responsible Party: Principal Investigator, David L Hare, Professor David L Hare, Austin Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H2006/02690; V1111-1166-3083 (Other: UTN)
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease; Atherosclerosis
Keywords: radial artery; right internal thoracic artery; saphenous vein; grafts; coronary bypass surgery
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis | interventions — Coronary Artery Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Other): Radial Artery versus Right Internal Thoracic Artery when used as a coronary conduit in patients undergoing multi-vessel coronary artery bypass grafting.
  Interventions: Procedure: Coronary artery bypass grafting
- Group 2 (Other): Radial Artery versus Saphenous Vein when used as a coronary conduit in patients undergoing multi-vessel coronary artery bypass grafting.
  Interventions: Procedure: Coronary artery bypass grafting

INTERVENTIONS:
Procedure: Coronary artery bypass grafting — Surgery performed due to coronary artery disease.

SUMMARY:
Coronary Artery Bypass Graft (CABG)Surgery is commonly used to treat patients with coronary artery disease (atherosclerosis) for the relief of angina (chest pain) and improve heart muscle function.

Healthy veins or arteries, referred to as 'conduits' from elsewhere in the patient's body, are grafted (attached) from the aorta to the coronary arteries, bypassing (via new routes) coronary artery narrowings caused by atherosclerosis (hardening of the arteries) and thereby improving the blood supply to the myocardium (heart muscle).

Over the years, a range of different veins and arteries from around the body have been used to bypass diseased coronary arteries. Typically, internal thoracic arteries from behind the breastbone and the saphenous veins from the legs are used for bypass. More recently, radial arteries from the forearm have also been used to bypass coronary arteries that are diseased (atherosclerotic). There is strong evidence to indicate that the left internal thoracic artery stays open the longest (i.e. has the highest patency) and achieves the best health outcomes. As a result, most cardiac surgeons use the left internal thoracic artery as their first choice of conduit (vessel used to bypass the blocked artery). However, many patients require multiple grafts and there is little evidence as to which grafts are the best conduits to use.

It has been suggested that the radial arteries might function better than saphenous veins as conduits. The Radial Artery Patency and Clinical Outcomes Trial(RAPCO) aims to compare patency of the radial arteries with the right internal thoracic artery and also with the saphenous vein.

DETAILED DESCRIPTION:
The Department of Cardiac Surgery at Austin Health is conducting a prospective randomised trial, stratified into two separate sub-studies. The first compares the radial artery with the right internal thoracic artery(as a free aorto-coronary graft) and the second comparies the radial artery with a saphenous vein graft. Each patient was to be followed for 10 years after their CABG surgery in order to assess both the pattern of graft survival over 10 years and also to record major clinical events.

The study was first given approval by the Austin Health Human Research Ethics Committee on August 18th,1995. Enrolment commenced in June 1996. Recruitment ceased in March 2005. Patients were randomly assigned to the control or experimental group, patients in both groups received the left internal thoracic artery to the left anterior decending(LAD) and the study graft as the second graft.

The gold standard measure for the comparison of conduits is through the use of post-operative angiograms. These angiograms assess how patent (open) the grafts are, and also offer quality assurance of the CABG surgery performed. To spread the graft patency end-points over the 10 years after CABG, patients undergo a second randomisation as to the time at which their graft patency is to be assessed. The timing of the graft study coronary angiogram is weighted towards the end of the 10 year period with the aim of having 10% at 1 year, 20% at 2 years, 20% at 5 years, 30% at 7.5 years and 30% at 10 years after CABG surgery. Clinical data is systematically collected to determine those patients who experience heart attack, repeat surgery, balloon angioplasty or death over subsequent years.

To enrich the number of mid-study graft patency end-points a protocol amendment(July 19th, 2002) was approved allowing patients to be offered a selective coronary angiogram at the 5 year anniversary of their surgery.

A further protocol amendment(November 16th, 2006) allowed coronary and graft CT angiography to be used optionally to replace selective angiography and also to offer all patients imaging at 10 years, in addition to the original pre-specified, randomised time of imaging.

As per the ethics approval and prior protocol amendments, lifelong followup is conducted on patients enrolled in the trial. As such, a RAPCO-Extension trial will be conducted, evaluating clinical outcomes at 15-years follow-up.

ELIGIBILITY:
Inclusion Criteria:

* The patient is scheduled for primary coronary artery bypass surgery alone ie. no reoperations, no associated procedures
* The patient requires more than 1 graft, that is, there are at least 2 coronary artery stenoses of > 70%.

Exclusion Criteria:

* Renal disease with a creatinine >0.30 mmol/L.
* Chronic heart failure (NYHA Class III or IV or ejection fraction <35% on angiography or radionuclide ventriculography).
* Associated major illnesses e.g., malignancy.
* Body mass index (BMI) > 35; weight (kg)/height(m2).
* Acute presentation, that is, those patients who have an acute myocardial infarct within one week prior to surgery or who present with cardiogenic shock.
* Technical exclusions e.g. sequential grafting.
* Failure to obtain informed consent.
* Off pump.

GROUP 1 Specific exclusions

* Failure to use radial artery due to abnormal Allen Test (>10 sec)
* Failure to be able to use the FRIMA eg. Chest trauma
* FEV1 < 50% of expected value
* Diabetic patients (IDDM or NIDDM) ≥60 years
* Patients ≥70 years

GROUP 2

* Specific exclusions
* Failure to use radial artery due to abnormal Allen Test (>10 sec)
* Failure to be able to use the saphenous vein eg. Varices, past trauma
* Diabetic patients <60 years of age
* Other patients <70 years of age

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605 (Estimated)
Dates: Start 1996-06; Primary Completion 2015-04 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Graft patency on all surviving trial patients. | Between 1-10 years from CABG surgery.
  Graft failure defined as either total occlusion, stenosis >80% or string sign.

SECONDARY OUTCOMES:
All cause mortality · | 10 years from CABG surgery
  Clinical follow-up and Australian National Death Registry
Event free Survival | 10 years from CABG surgery
  Events defined as all-cause mortality, myocardial infarction, revascularisation (percutaneous or surgical).

OTHER OUTCOMES:
[RAPCO-Extension trial] All cause mortality | 15 years from CABG Surgery
  Clinical follow-up
[RAPCO-Extension trial] Event free survival | 15 years from CABG surgery
  Events defined as all-cause mortality, myocardial infarction, revascularisation (adjudication of all events)
[RAPCO-Extension trial] Myocardial infarction | 15 years from CABG surgery
  Rates of myocardial infarction (adjudication according to the fourth universal definition of MI)
[RAPCO-Extension trial] Revascularisation | 15 years from CABG surgery
  Rates of coronary revascularisation (either PCI or redo-CABG)

CONTACTS AND LOCATIONS:
Overall Officials: David L Hare, MB BS DPM FRACP FESC FACC, Study Director — Austin Health
Locations (1):
- Austin Health, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buxton BF, Hayward PA, Raman J, Moten SC, Rosalion A, Gordon I, Seevanayagam S, Matalanis G, Benedetto U, Gaudino M, Hare DL; RAPCO Investigators*. Long-Term Results of the RAPCO Trials. Circulation. 2020 Oct 6;142(14):1330-1338. doi: 10.1161/CIRCULATIONAHA.119.045427. Epub 2020 Oct 5. PMID 33017209